CLINICAL TRIAL: NCT06493838
Title: Clinical Efficacy of Prophylactic Intravenous Neostigmine and Atropine in Preventing Post-Dural Puncture Headache Among Parturient Undergoing Spinal Anesthesia for Cesarean Section: A Double-blind Randomized Placebo-controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Ass professor anesthesia and pain, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0379/2023
Record Dates: First submitted 2024-06-30; First posted 2024-07-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Neostigmine; Atropine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): intravenous 50 mL of sterile saline 0.9% injection of 0.9% after umbilical cord clamping.
  Interventions: Drug: intravenous 50 mL of saline injection of 0.9% after umbilical cord clamping.
- Neostgmine group (Active Comparator): Neostigmine 20μg/kg (Neostigmine Methylsulphate 0.5 mg, Amriya Pharm.Ind.) and atropine 0.01 mg/kg (diluted in 50 ml saline; 0.9% for 10 min) following umbilical cord clamping.
  Interventions: Drug: Neostigmine 20μg/kg (Neostigmine Methylsulphate 0.5 mg, Amriya Pharm.Ind.) and atropine 0.01 mg/kg (diluted in 50 ml saline; 0.9% for 10 min) following umbilical cord clamping.

INTERVENTIONS:
Drug: intravenous 50 mL of saline injection of 0.9% after umbilical cord clamping. — intravenous 50 mL of saline injection of 0.9% after umbilical cord clamping.
  Arms: Control group
Drug: Neostigmine 20μg/kg (Neostigmine Methylsulphate 0.5 mg, Amriya Pharm.Ind.) and atropine 0.01 mg/kg (diluted in 50 ml saline; 0.9% for 10 min) following umbilical cord clamping. — Neostigmine 20μg/kg (Neostigmine Methylsulphate 0.5 mg, Amriya Pharm.Ind.) and atropine 0.01 mg/kg (diluted in 50 ml saline; 0.9% for 10 min) following umbilical cord clamping.
  Arms: Neostgmine group

SUMMARY:
Post dural puncture headache is a distressing issue, many measures tried to treat symptoms but few delt with prevention.

ELIGIBILITY:
Inclusion Criteria:

* Parturient ladies
* Age ranges from 18 to 35 years old.
* ASA II with elective caesarean section under sub-arachnoid block

Exclusion Criteria:

* BMI >35
* Refusal to participate
* surgical complications necessitating a blood transfusion
* Emergency caesarean section
* the need for endotracheal intubation or vasopressors
* any contraindication to regional anesthesia (such as a history of persistent cephalgia, convulsions, cerebrovascular events

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — We target obstetric population
Enrollment: 180 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients with post dural puncture headache | first 5 days post-partum
  Number of patients develop post dural puncture headache

SECONDARY OUTCOMES:
Severity of post dural puncture headache | first 5 days post-partum
  Visual analogue scale score for pain assessment. from 0 to ten. 0= no pain 1-3= mild pain....4-6= moderate pain ... 7-10= severe pain
onset and duration of post dural puncture headache | 5 days post partum
  Time when visual analogue scale score increase and duration until return to 0. Visual analogue scale score for pain assessment. from 0 to ten. 0= no pain 1-3= mild pain....4-6= moderate pain ... 7-10= severe pain
Analgesic request | 24 hours after operation
  First time to analgesic request from block
Analgesc requirements | 2 days after operation
  Total analgesic requirements
frequency of analgesic doses | 5 days
  number of analgesic doses given to the patient
incidence of complications related to the procedure | 6 hours after procedure
  number of patients with adverse events as bradycardia, tachcardia, miosis,muscle cramps, twitches, colics, hypotension